CLINICAL TRIAL: NCT02052804
Title: Understanding and Treating Heart Failure With Preserved Ejection Fraction: Novel Mechanisms, Diagnostics and Potential Therapeutics
Acronym: Alberta HEART
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Justin Ezekowitz, Associate Professor, University of Alberta; Director, Heart Function Clinic- Mazankowski Alberta Heart Institute, University of Alberta
Other Study IDs: AHFMRITG200801018
Record Dates: First submitted 2014-01-21; First posted 2014-02-03 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of this study are: 1) to design new diagnostic criteria used to accurately define heart failure with preserved ejection fraction (HFpEF); 2) to better define the risk factors associated with HFpEF; 3) to elucidate the clinical, cellular and molecular mechanisms involved with the development and progression of HFpEF; 4) to design and test new therapeutic strategies for patients with HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 No clinically overt heart failure
* Group 2 Known coronary artery disease
* Group 3 Known heart failure with preserved ejection fraction
* Group 4 Known heart failure with reduced ejection fraction
* Group 5 Healthy age-matched controls

Exclusion Criteria:

* Age <18 years
* Known malignancy with expected survival <1 year
* Pregnant or recent pregnancy <6 months
* Recent event (<2 weeks since Acute Coronary Syndrome, Heart failure or other admission
* Severe mitral or aortic stenosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Alberta, Canada with heart failure or at risk for developing heart failure
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2009-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Percent of patients meeting new diagnostic criteria for HFpEF | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Dyck, PhD, Study Director — University of Alberta
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

REFERENCES:
- [Derived] Zordoky BN, Sung MM, Ezekowitz J, Mandal R, Han B, Bjorndahl TC, Bouatra S, Anderson T, Oudit GY, Wishart DS, Dyck JR; Alberta HEART. Metabolomic fingerprint of heart failure with preserved ejection fraction. PLoS One. 2015 May 26;10(5):e0124844. doi: 10.1371/journal.pone.0124844. eCollection 2015. PMID 26010610
- [Derived] Ezekowitz JA, Becher H, Belenkie I, Clark AM, Duff HJ, Friedrich MG, Haykowsky MJ, Howlett JG, Kassiri Z, Kaul P, Kim DH, Knudtson ML, Light PE, Lopaschuk GD, McAlister FA, Noga ML, Oudit GY, Paterson DI, Quan H, Schulz R, Thompson RB, Weeks SG, Anderson TJ, Dyck JR. The Alberta Heart Failure Etiology and Analysis Research Team (HEART) study. BMC Cardiovasc Disord. 2014 Jul 25;14:91. doi: 10.1186/1471-2261-14-91. PMID 25063541